CLINICAL TRIAL: NCT02144090
Title: Opsens Optowire for Fractional Flow Reserve - The O2 Pilot Study
Acronym: O2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Opsens, Inc. (Industry); International Chair on Interventional Cardiology and Transradial Approach (Other)
Responsible Party: Principal Investigator, Olivier F. Bertrand, Study Principal Investigator, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: O2 Pilot Study
Record Dates: First submitted 2014-05-15; First posted 2014-05-21 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Stable Angina; Unstable Angina Pectoris; Chest Pain; Ischemia
Keywords: Angiography; Angioplasty; Coronary artery disease; Diagnostic; Fractional flow reserve
MeSH Terms: conditions — Angina, Stable; Angina, Unstable; Chest Pain; Ischemia; Coronary Artery Disease; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fractional flow reserve (Experimental): Fractional flow reserve measurement
  Interventions: Device: Fractional flow reserve measurement

INTERVENTIONS:
Device: Fractional flow reserve measurement — Fractional flow reserve measurement
  Other Names: Opsens Optowire and Optomonitor

SUMMARY:
The purpose of this study is to assess the usability and safety of the Opsens OptoWire and Optomonitor in measuring fractional flow reserve (FFR) in patients with coronary artery disease who are undergoing a coronary angiogram.

DETAILED DESCRIPTION:
Fractional flow reserve (FFR) measurement involves determining the ratio between the maximum achievable blood flow in a diseased coronary artery and the theoretical maximum flow in a normal coronary artery. An FFR of 1.0 is widely accepted as normal. An FFR value lower than 0.75 - 0.80 is generally considered to be associated with myocardial ischemia (MI).

FFR is easily measured during routine coronary angiography by using a pressure wire to calculate the ratio between coronary pressure distal to a coronary artery stenosis and aortic pressure under conditions of maximum myocardial hyperemia. This ratio represents the potential decrease in coronary flow distal to the coronary stenosis.

Over the past decade, FFR measurement has been increasingly used in cardiac catheterization laboratories. It provides a quantitative assessment of the functional severity of a coronary artery stenosis identified during coronary angiography and cardiac catheterization.

Opsens, Inc. has developed a new pressure wire for use in determining FFR in coronary arteries; the OptoWire. The OptoWire is an instrumented guide wire with a fiber optic pressure sensor mounted 3.5 cm proximal to the tip. The Optowire measures blood pressure during diagnostic and/or interventional procedures when used in combination with the OptoMonitor.

The O2 study is a pilot study which aims to provide preliminary experience in human patients with coronary artery disease. The study data will also be used as part of design validation.

The O2 study is a prospective single arm study designed to assess the usability, functionality, and safety of the Optowire and Optomonitor in patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with

  * Stable angina or,
  * Unstable angina pectoris or,
  * Atypical chest pain or no chest pain but with suspected ischemia
* At least one moderate lesion in native coronary artery thought to produce ischemia
* Operator and patient agree for procedures
* Patient (> 18 years) has signed a written informed consent prior to procedure

Exclusion Criteria:

* Lesions with angiographic 'haziness' or suspected to contain thrombus
* Post-coronary artery bypass grafting
* Total occlusion
* If use of atherectomy device is indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Safety and handling assessment of the Optowire | Patients will be followed through removal of the OptoWire from percutaneous insertion site and completion of the cardiac catheterization procedure (expected average <1hr)
  1. Safely reach and cross a target lesion;
  2. perform an FFR measurement using the Optowire and Optomonitor according to the product user guide;
  3. disconnect the proximal connector on the OptoWire during the procedure, placing an interventional device (if necessary), and reconnecting the Optowire proximal connector;
  4. safely remove the Optowire from the coronary artery.
  Dedicated questionnaires will be used for such assessment

SECONDARY OUTCOMES:
Comparison of FFR values measured with Optowire vs. with FFR guide wire used in standard practice | Patients will be followed through removal of the OptoWire from percutaneous insertion site and completion of the cardiac catheterization procedure (expected average <1hr)
  In selected cases, the operator may choose to perform FFR measurements using currently approved FFR wires. Values obtained with standard FFR wires and Optowire may therefore be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier F Bertrand, MD PhD, Principal Investigator — International Chair on Interventional Cardiology and Transradial Approach
Locations (1):
- IUCPQ - Laval Hospital, Québec, Quebec, Canada